CLINICAL TRIAL: NCT05497388
Title: Efficacy of Serious Game Interventions on Hepatitis C Education for HIV-Positive Men Who Have Sex With Men: A Randomized Controlled Trial
Brief Title: Efficacy of Serious Game Interventions on HCV Education for HIV Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202206084RIND
Record Dates: First submitted 2022-07-28; First posted 2022-08-11 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: MSM; Hepatitis C; Health Belief Patterns; Serious Games
MeSH Terms: conditions — HIV Infections; Hepatitis C

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web for HCV education (No Intervention)
- Serious Game for HCV education (Experimental)
  Interventions: Other: Serious Game

INTERVENTIONS:
Other: Serious Game — using Serious Game for HCV education
  Arms: Serious Game for HCV education

SUMMARY:
Hepatitis C transmission has a high rate of infection and re-infection among PLWH men who have sex with men (MSM), and co-infection increases liver and HIV morbidity.

The MSM group has a low level of awareness and perception of hepatitis C, and lacks health beliefs and prevention behaviors about hepatitis C. In the absence of hepatitis C cognition and health belief, it should be possible to use the health belief model to intervene and design teaching programs to improve the effectiveness of hepatitis C prevention and treatment. In the past, hepatitis C prevention education mostly focused on people who inject drugs (PWID), and was taught in traditional teaching methods. However, the common cause of hepatitis C infection among drug addicts is the sharing of needles and equipment. Education is mainly based on drug harm reduction and prevention education, while the MSM group is infected with hepatitis C mainly through risky sexual behaviors. The hepatitis C prevention education of drug addicts is adopted The content is clearly not applicable to the MSM population. Due to the stigma of PLWH's MSM in the society, individual cases will be subject to prejudice, discrimination and unfair treatment, and they are worried about being excluded from outsiders. Therefore, it is necessary to provide a learning environment with a sense of privacy, security and respect.

Serious Games is an educational game that provides a ubiquitous way of learning, using smartphones as a teaching tool, allowing learners to maintain a sense of privacy. Positive outcomes in cognitions, attitudes and behaviours related to health promotion and disease management. In terms of sexually transmitted diseases prevention measures, game content can be formulated for specific ethnic groups, and sensitive topics can be placed in the game. Without being exposed to real risks, players can simulate the consequences of various risks and corresponding prevention methods to prevent Motivate learners to solve problems and learn motivation, and give clear feedback, thereby increasing the knowledge of hepatitis C, health beliefs and the effectiveness of preventive self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected men who have sex with men aged 20-45
* Can communicate in appropriate language and understand the research content
* Able to use smartphone products

Exclusion Criteria:

* Unable to fully participate in this study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The effect of "serious game-assisted teaching" intervention program on MSM. | 12 weeks after intervention.
  The changes of Questionnaire score of hepatitis C knowledge, health beliefs, and self-efficacy will be measured, Questionnaire including:
  1. HCV Knowledge Scale:Scores range from 0 to 15, with higher scores representing higher knowledge of hepatitis C
  2. Health Belief Model (HBM):Scores range from 1 to 28, with higher scores representing more positive hepatitis C prevention beliefs.
  3. Self-Efficacy Scale:Scores range from 1 to 8, with higher scores representing better self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Yi Ting Chen, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No